CLINICAL TRIAL: NCT04868110
Title: Preventing Excessive Weight Gain and Maternal and Infant Fat Accretion by Increasing Fiber Intake and Changing the Maternal Microbiome During Pregnancy
Brief Title: Preventing Excessive Weight Gain and Maternal and Infant Fat Accretion
Acronym: SPROUT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00145397
Record Dates: First submitted 2021-04-14; First posted 2021-04-30 (Actual); Results first posted 2025-01-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2024-12

CONDITIONS: Gestational Weight Gain; Maternal Fat Accretion; Infant Fat Accretion
Keywords: Fat mass; Gestational weight gain; Infant fat mass; High fiber; Microbiome
MeSH Terms: conditions — Gestational Weight Gain

STUDY DESIGN:
Intervention Model Description: Women in the control group will participate in weekly lessons for 18 weeks on eating a high fiber diet and will received daily snacks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): Women in the usual care group, will received standard care from the obstetrician.
- High fiber (Experimental): Women in high fiber group will receive education on consuming a high fiber diet, including weekly lessons and daily snacks.
  Interventions: Behavioral: High fiber diet

INTERVENTIONS:
Behavioral: High fiber diet — A registered dietitian will delivered the lessons on consuming a high fiber diet to small groups to increased engage and material retention. These lessons will last 18 weeks.
  Arms: High fiber

SUMMARY:
The purpose of this study is to learn if consuming a high fiber diet will reduce gestational weight gain and maternal and infant fat accretion.

ELIGIBILITY:
Inclusion Criteria:

* Pre-pregnancy BMI 18.5 - 45.0 kg/m2

Exclusion Criteria:

* Comsuming more than 20 g/day of fiber
* No phone and internet access
* Pre-gestational diabetes
* Diagnosed with diabetes
* Pre-eclampsia
* Hypertension
* Other metabolic abnormalities
* Asthma
* Heart disease
* Smoking
* Drug abuse
* Recent antibiotic use
* Pregnancies of multiples

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2021-06-28 (Actual); Primary Completion 2023-09-29 (Actual); Study Completion 2023-10-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Holly Hull, PhD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- The University of Kansas Medical Center, Kansas City, Kansas, United States

REFERENCES:
- [Derived] Herman A, Hand LK, Gajewski B, Krase K, Sullivan DK, Goetz J, Hull HR. A high fiber diet intervention during pregnancy: The SPROUT (Single goal in PRegnancy to optimize OUTcomes) protocol paper. Contemp Clin Trials. 2024 Feb;137:107420. doi: 10.1016/j.cct.2023.107420. Epub 2023 Dec 23. PMID 38145714

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Usual Care | High Fiber
Started | 26 | 25
Completed | 23 | 21
Not Completed | 3 | 4
Not completed — Withdrawal by Subject | 3 | 4

BASELINE CHARACTERISTICS:
Population: Three participants withdrew from the study after enrolling, but prior to the baseline visit.
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | High Fiber | Total
Number analyzed (Participants) | 24 | 24 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 24 | 24 | 48
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.92 (4.86) | 29.79 (4.62) | 30.85 (4.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 24 | 48
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 4 | 6
  Not Hispanic or Latino | 22 | 20 | 42
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 19 | 18 | 37
  More than one race | 3 | 2 | 5
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 24 | 24 | 48
Pre-pregnancy Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 26.33 (4.95) | 24.92 (4.03) | 25.62 (4.52)

OUTCOME MEASURES:

1. Primary Outcome: Maternal Weight Changes
Description: Assess weight change between groups
Time Frame: Baseline through 2-mounths postpartum
Population: Thirteen participants were removed from the analysis due to a diagnosis of gestational hypertension or hypertensive disorder of pregnancy.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Usual Care | High Fiber
Number analyzed (Participants) | 15 | 16
kg
  Weight at Baseline (kg) | 70.20 (10.44) | 66.47 (7.04)
  Weight at End of Pregnancy (kg) | 80.12 (10.00) | 75.80 (6.89)
  Weight at 2mo postpartum (kg) | 73.53 (10.04) | 67.99 (7.36)

2. Primary Outcome: Maternal Fat Accretion Changes
Description: Assess fat accretion change between groups using the Selinger four-compartment model
Time Frame: Baseline through 2-mounths postpartum
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent fat mass
Arm/Group | Usual Care | High Fiber
Number analyzed (Participants) | 15 | 16
percent fat mass
  Percent Fat Mass at Baseline | 33.49 (5.96) | 32.27 (5.18)
  Percent Fat Mass at End of Pregnancy | 36.74 (5.05) | 34.91 (4.33)
  Percent Fat Mass at 2mo postpartum | 36.35 (5.95) | 34.38 (5.65)

3. Primary Outcome: Identify Changes in Fiber Intake
Description: Compare fiber intake between groups by using 24-hour dietary recalls
Time Frame: Baseline through 2-months postpartum
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: g/day
Arm/Group | Usual Care | High Fiber
Number analyzed (Participants) | 15 | 16
g/day
  Total Dietary Fiber Intake at Baseline (g/day) | 19.01 (3.88) | 21.84 (7.51)
  Total Dietary Fiber Intake at End of Pregnancy (g/day) | 19.35 (8.05) | 35.09 (7.37)
  Total Dietary Fiber Intake at 2mo postpartum (g/day) | 19.62 (6.78) | 29.71 (10.63)

4. Primary Outcome: Identify Changes in Dietary Quality
Description: Compare dietary quality between groups using the Alternative Healthy Eating Index (AHEI) scoring ranges from 0 to 100 (higher score means a better diet quality).
Time Frame: Baseline through 2-months postpartum
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: AHEI score
Arm/Group | Usual Care | High Fiber
Number analyzed (Participants) | 15 | 16
AHEI score
  Alternative Healthy Eating Index (AHEI) Total Score at Baseline | 54.59 (9.82) | 62.51 (10.95)
  Alternative Healthy Eating Index (AHEI) Total Score at End of Pregnancy | 50.06 (11.34) | 70.12 (12.41)
  Alternative Healthy Eating Index (AHEI) Total Score at 2mo postpartum | 51.43 (10.34) | 62.53 (9.33)

5. Secondary Outcome: Infant Fat Accrual
Description: Identify differences in early infant fat accrual between group by completing body composition measurements including but not limited to Dual energy x-ray absorptiometry (DXA) and PeaPod
Time Frame: Birth to 12-month old
Population: Of the participants that completed the 2-week and 12-month visits, many refused or were uncooperative during the DXA scan. And even a higher percentage were deemed unusable scans due to infant movement.
Measure: Mean (Standard Deviation); unit: percent fat mass
Arm/Group | Usual Care | High Fiber
Number analyzed (Participants) | 10 | 11
percent fat mass
  Percent Fat Mass at 2-weeks | 17.20 (2.52) | 17.26 (3.23)
  Percent Fat Mass at 12-months | 34.89 (3.16) | 32.62 (3.57)

6. Secondary Outcome: Maternal Weight
Description: Assess weight change
Time Frame: 2-months through 12-months postpartum
Population: Between the 2mo and 12mo timepoint, one participant withdrew from high fiber group of the study (Baseline to 2mo postpartum, Usual care: 15, High Fiber:16).
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Usual Care | High Fiber
Number analyzed (Participants) | 15 | 15
kg
  Weight at 6mo postpartum (kg) | 71.67 (11.87) | 65.53 (8.07)
  Weight at 12mo postpartum (kg) | 71.65 (11.56) | 64.58 (8.30)

7. Secondary Outcome: Maternal Fat Accretion
Description: Assess fat accretion change between groups using the Selinger four-compartment model
Time Frame: 2-months through 12-months postpartum
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: percent fat mass
Arm/Group | Usual Care | High Fiber
Number analyzed (Participants) | 15 | 15
percent fat mass
  Percent Fat Mass at 6mo postpartum | 34.79 (8.19) | 30.92 (5.28)
  Percent Fat Mass at 12mo postpartum | 33.69 (9.09) | 30.81 (6.76)

8. Secondary Outcome: Dietary Fiber Intake
Description: Assess differences using 24h recalls
Time Frame: 2-months through 12-months postpartum
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: g/day
Arm/Group | Usual Care | High Fiber
Number analyzed (Participants) | 15 | 15
g/day
  Total Dietary Fiber Intake at 6mo postpartum | 19.48 (6.72) | 26.94 (7.58)
  Total Dietary Fiber Intake at 12mo postpartum | 17.87 (6.31) | 23.80 (7.13)

9. Secondary Outcome: Dietary Quality
Description: as for outcome 4
Time Frame: 2-months through 12-months postpartum
Population: Between the 2mo and 12mo timepoint, one participant withdrew from the study
Measure: Mean (Standard Deviation); unit: AHEI score
Arm/Group | Usual Care | High Fiber
Number analyzed (Participants) | 15 | 15
AHEI score
  Alternative Healthy Eating Index (AHEI) Total Score at 6mo postpartum | 49.47 (11.72) | 66.05 (13.69)
  Alternative Healthy Eating Index (AHEI) Total Score at 12mo postpartum | 48.66 (12.14) | 61.59 (10.11)

ADVERSE EVENTS:
Time Frame: Adverse event data was tracked and monitored from baseline (12-20 weeks gestation) until 30 days post invention (up to 2 weeks postpartum).
Arm/Group | Usual Care | High Fiber
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 0/24 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-01-12): https://cdn.clinicaltrials.gov/large-docs/10/NCT04868110/Prot_SAP_000.pdf
  • Informed Consent Form (2022-01-12): https://cdn.clinicaltrials.gov/large-docs/10/NCT04868110/ICF_001.pdf